CLINICAL TRIAL: NCT01994746
Title: Efficacy and Safety of Nasal Glucagon for Treatment of Insulin Induced Hypoglycemia in Adults With Diabetes
Brief Title: Efficacy and Safety of Nasal Glucagon for Treatment of Hypoglycemia in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Collaborators: T1D Exchange Clinic Network Coordinating Center (Unknown); Locemia Solutions ULC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 16422; INGluc001 (Other: Jaeb Center for Health Research); I8R-MC-IGBC (Other: Eli Lilly and Company); AMG106 (Other: Locemia)
Record Dates: First submitted 2013-11-20; First posted 2013-11-26 (Estimated); Results first posted 2016-10-10 (Estimated); Last update posted 2019-09-23 (Actual); Status verified 2019-09

CONDITIONS: Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nasal Glucagon (Experimental): At one visit, a glucagon dose of 3 mg was administered in a nostril with a prefilled delivery device that delivers a single dose upon activation.
  Interventions: Drug: Nasal Glucagon
- Intramuscular Glucagon (Active Comparator): At a separate visit, 1 mg of glucagon was administered into the deltoid muscle of the non-dominant arm (intramuscular [IM]).
  Interventions: Drug: Intramuscular Glucagon

INTERVENTIONS:
Drug: Nasal Glucagon
  Other Names: AMG504-1; LY900018
  Arms: Nasal Glucagon
Drug: Intramuscular Glucagon
  Other Names: GlucaGen HypoKit
  Arms: Intramuscular Glucagon

SUMMARY:
The purpose of this study is to assess the efficacy, pharmacokinetics (PK), pharmacodynamics (PD), and safety of 3 milligrams (mg) glucagon (glucagon nasal powder) administered nasally compared with commercially available glucagon given by intramuscular injection.

DETAILED DESCRIPTION:
Each glucagon dosing visit was conducted after an overnight fast of at least 8 h with a starting plasma glucose >= 90 mg/dL. Hypoglycemia was induced by an intravenous (IV) infusion of regular insulin diluted in normal saline during the clinic visit. Five minutes after stopping the insulin infusion (once the plasma glucose was <60 mg/dL), participants were treated with either a 3 mg glucagon dose nasally or 1 mg of glucagon administered by intramuscular (IM) injection.

After a wash-out period of 7 days or more, participants returned to the clinic and the procedure repeated with each participant crossed over to the other treatment. As such, each participant underwent two episodes of insulin-induced hypoglycemia in random order and received glucagon nasal powder during one episode and commercially available glucagon (GlucaGen, Novo Nordisk) by IM injection during the other episode.

ELIGIBILITY:
Inclusion Criteria:

To be eligible, the following inclusion criteria must be met:

* Clinical diagnosis of either type 1 diabetes receiving daily insulin since the time of diagnosis for at least 2 years or type 2 diabetes receiving multiple daily insulin doses for at least 2 years
* At least 18.0 years of age and less than 65.0 years
* Body mass index (BMI) greater than or equal to 20.0 and below or equal to 35.0 kilograms per meter squared (kg/m²)
* Weighs at least 50 kg (110 pounds)
* Females must meet one of the following criteria:

  * Of childbearing potential but agree to use an accepted contraceptive regimen as described in the study procedure manual throughout the entire duration of the study (from the screening until study completion)
  * Of non-childbearing potential, defined as a female who has had a hysterectomy or tubal ligation, is clinically considered infertile or is in a menopausal state (at least 1 year without menses)
* In good general health with no conditions that could influence the outcome of the trial, and in the judgment of the Investigator is a good candidate for the study based on review of available medical history, physical examination and clinical laboratory evaluations
* Willingness to adhere to the study requirements

Exclusion Criteria:

An individual is not eligible if any of the following exclusion criteria are present:

* Females who are pregnant according to a positive urine pregnancy test, actively attempting to get pregnant, or are lactating
* History of hypersensitivity to glucagon or any related products or severe hypersensitivity reactions (such as angioedema) to any drugs
* Presence of cardiovascular, gastrointestinal, liver or kidney disease, or any other conditions which in the judgment of the investigator could interfere with the absorption, distribution, metabolism or excretion of drugs or could potentiate or predispose to undesired effects
* History of pheochromocytoma (i.e. adrenal gland tumor) or insulinoma.
* History of an episode of severe hypoglycemia (as defined by an episode that required third party assistance for treatment) in the 1 month prior to enrolling in the study
* Use of daily systemic beta-blocker, indomethacin, warfarin or anticholinergic drugs
* History of epilepsy or seizure disorder
* Regularly consumes 3 or more alcoholic beverages per day
* Use of an Investigational Product in another clinical trial within the past 30 days
* Donated 225 milliliters (mL) or more of blood in the previous 8 weeks before the first glucagon dosing

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 77 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (8):
- United States (8):
  - Barbara Davis Center for Diabetes, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - University of Florida, Gainesville, Florida
  - Riley Hospital for Children Indiana University Health, Indianapolis, Indiana
  - University of Minnesota, Minneapolis, Minnesota
  - UPA Buffalo, Buffalo, New York
  - Oregon Health and Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and EU, whichever is later. Data will be indefinitely available for requesting.
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: https://vivli.org/

REFERENCES:
- [Background] Rickels MR, Ruedy KJ, Foster NC, Piche CA, Dulude H, Sherr JL, Tamborlane WV, Bethin KE, DiMeglio LA, Wadwa RP, Ahmann AJ, Haller MJ, Nathan BM, Marcovina SM, Rampakakis E, Meng L, Beck RW; T1D Exchange Intranasal Glucagon Investigators. Intranasal Glucagon for Treatment of Insulin-Induced Hypoglycemia in Adults With Type 1 Diabetes: A Randomized Crossover Noninferiority Study. Diabetes Care. 2016 Feb;39(2):264-70. doi: 10.2337/dc15-1498. Epub 2015 Dec 17. PMID 26681725
- [Derived] Seaquist E, Gimenez M, Yan Y, Matsuhisa M, Kao CY, Wadwa RP, Nagai Y, Khunti K. Nasal Glucagon Reverses Insulin-induced Hypoglycemia With Less Rebound Hyperglycemia: Pooled Analysis of Clinical Trials. J Endocr Soc. 2024 Feb 26;8(4):bvae034. doi: 10.1210/jendso/bvae034. eCollection 2024 Feb 19. PMID 38444629

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 77 Type 1 (T1D) and 6 Type 2 diabetes (T2D) participants were recruited. Results reported include T1D participants only since this was the pre-specified primary population.
Groups:
- NG 1st/IM Glucagon 2nd: At the first visit, 3 milligrams (mg) of nasal glucagon (NG). At the second visit, 1 mg of intramuscular (IM) glucagon.
- IM Glucagon 1st/NG 2nd: At the first visit, 1 mg of IM glucagon. At the second visit, 3 mg of NG glucagon.
Period: First Visit
Arm/Group | NG 1st/IM Glucagon 2nd | IM Glucagon 1st/NG 2nd
Started | 39 | 38
Received At Least 1 Dose | 39 | 38
Completed | 39 | 38
Not Completed | 0 | 0
Period: Second Visit
Arm/Group | NG 1st/IM Glucagon 2nd | IM Glucagon 1st/NG 2nd
Started | 38 (One participant requested to withdraw after completing the first dosing visit.) | 38
Completed Both Dosing Visits | 38 | 38
Completed | 38 | 38
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Participants that received at least one does of study drug.
Groups:
- All Study Participants: At one visit, a nasal glucagon (NG) dose of 3 mg. At another visit, 1 mg intramuscular (IM) glucagon The order of the visits were randomized.
Arm/Group | All Study Participants
Number analyzed (Participants) | 77
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 77
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 33 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 75
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 74
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77

OUTCOME MEASURES:

1. Primary Outcome: Increase in Plasma Glucose Level to >=70mg/dL or an Increase of >=20mg/dL From Glucose Nadir
Description: Increase in blood glucose to ≥70 mg/dL or an increase of ≥20 mg/dL from glucose nadir within 30 minutes after receiving study glucagon, without receiving additional actions to increase the blood glucose level defines treatment success. Due to the residual activity of circulating insulin, glucose nadir was defined as the minimum glucose measurement at the time of, or within 10 minutes following glucagon administration.
Time Frame: Within 30 minutes after receiving glucagon at both dosing visits (glucose was measured at pre-dose; 5, 10, 15, 20, 25, and 30 minutes following glucagon administration)
Population: All enrolled participants who completed both eligible Study/Dosing Visits.
Measure: Number; unit: percentage of participants
Groups:
- Nasal Glucagon (NG): At one visit, 3 mg of NG.
- Intramuscular (IM) Glucagon: At a separate visit, 1 mg of IM glucagon.
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
percentage of participants | 98.7 | 100

2. Secondary Outcome: Nasal and Non-nasal Effects/Symptoms
Description: Symptoms of runny nose, nasal congestion and/or itching, sneezing, watery and/or itchy eyes, redness of eyes, and itching of ears and/or throat were assessed. This was done via the "Nasal Non-nasal Score Questionnaire". Each of the 9 symptoms is assigned an integer value from 0 to 3; higher values indicate more severe symptoms (a score of 0 indicates no symptoms). The reported results indicate the cohort median out of a possible maximum value of 27 (summing all 9 questions for each subject and reporting the median/IQR across participants).
Time Frame: Pre-dose; 15, 30, 60, and 90 post glucagon administration
Population: All enrolled T1D participants that completed the required dosing visits. Study dosing visits occur on Day 0 and then again after the washout period between Day 7 to Day 28.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 77 | 76
units on a scale
  Pre-dose | 0.00 [0.00 to 1.00] | 0.00 [0.00 to 1.00]
  15 minutes post glucagon administration | 2.00 [1.00 to 5.00] | 0.00 [0.00 to 0.00]
  30 minutes post glucagon administration | 1.00 [0.00 to 3.00] | 0.00 [0.00 to 0.50]
  60 minutes post glucagon administration | 1.00 [0.00 to 3.00] | 0.00 [0.00 to 0.00]
  90 minutes post glucagon administration | 1.00 [0.00 to 2.50] | 0.00 [0.00 to 0.00]

3. Secondary Outcome: Recovery From Symptoms of Hypoglycemia
Description: Recovery from hypoglycemia symptoms were assessed using the Edinburgh Hypoglycemia Scale. The Edinburgh Hypoglycemia Symptom Scale measures the intensity of 15 commonly experienced hypoglycemic symptoms on a 7-point Likert scale (1 = not present, 7 = very intense). The higher the score, the more intense the hypoglycemia symptoms. The sum of each symptom score would yield a range of 15 to 105 (i.e., 15 x 7 =105). The total score was calculated as the sum of each symptom score minus 15, and summarized at each time point by treatment group.
Time Frame: Pre-dose;15, 30, 45 and 60 minutes following administration of glucagon
Population: All enrolled participants who completed at least one post administration survey.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 77 | 76
units on a scale
  Pre-dose | 8.0 (7.7) | 7.8 (7.1)
  15 minutes post glucagon administration | 8.8 (8.3) | 5.3 (5.2)
  30 minutes post glucagon administration | 4.9 (4.7) | 3.5 (3.9)
  45 minutes post glucagon administration | 3.8 (3.1) | 3.0 (3.0)
  60 minutes post glucagon administration | 3.9 (3.1) | 3.1 (2.9)

4. Secondary Outcome: Time From Glucagon Administration to Blood Glucose >/=70 mg/dL or an Increase ≥20 mg/dL in Blood Glucose From Nadir
Description: The mean time from glucagon administration to blood glucose >/=70 mg/dL or an increase ≥20 mg/dL in blood glucose from nadir.
Time Frame: Pre-dose; 5, 10, 15, 20, 25, and 30 minutes following glucagon administration
Population: All enrolled participants that completed the required dosing visits with eligible glucose and glucagon levels. Study dosing visits occur on Day 0 and then again after the washout period between Day 7 to Day 28.
Measure: Number; unit: minutes
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
minutes | 16.2 | 12.2

5. Secondary Outcome: Area Under the Curve From Time Zero to the Last Quantifiable Concentration (AUC0-t) of Baseline-Adjusted Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: All enrolled participants that completed the required dosing visits with available pharmacokinetics (PK) data. Study dosing visits occurred on Day 0 and then again after the washout period between Day 7 to Day 28.
Measure: Mean (Standard Deviation); unit: hour*picograms per milliliter (hr*pg/mL)
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
hour*picograms per milliliter (hr*pg/mL) | 1882.48 (1216.27) | 2521.87 (971.07)

6. Secondary Outcome: Maximum Change From Baseline Concentration (Cmax) of Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: picograms per milliliter (pg/mL)
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
picograms per milliliter (pg/mL) | 3025.37 (1981.62) | 3553.43 (1746.66)

7. Secondary Outcome: Time to Maximum Change From Baseline Concentration (Tmax) of Glucagon
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: as for outcome 5
Measure: Median (Full Range); unit: hours
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
hours | 0.33 [0.17 to 1.50] | 0.25 [0.08 to 1.00]

8. Secondary Outcome: Area Under the Effect Concentration Time Curve (AUEC0-1.5) of Baseline-Adjusted Glucose From Time Zero up to 90 Minutes
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: All enrolled participants that completed the required dosing visits with available pharmacodynamics (PD) data. Study dosing visits occurred on Day 0 and then again after the washout period between Day 7 to Day 28.
Measure: Mean (Standard Deviation); unit: hr*mg/dL
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
hr*mg/dL | 106.39 (42.60) | 124.47 (38.95)

9. Secondary Outcome: Maximum Change From Baseline Concentration (Cmax) of Glucose
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: milligrams per deciliter (mg/dL)
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
milligrams per deciliter (mg/dL) | 114.80 (47.45) | 130.72 (44.15)

10. Secondary Outcome: Time to Maximum Change From Baseline Concentration (Tmax) of Glucose
Time Frame: Pre-dose; 5, 10, 15, 20, 25, 30, 40, 50, 60 and 90 minutes following glucagon administration
Population: as for outcome 8
Measure: Median (Full Range); unit: hours
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Number analyzed (Participants) | 75 | 75
hours | 1.5 [0.5 to 1.5] | 1.5 [0.5 to 1.5]

ADVERSE EVENTS:
Time Frame: Through study completion, up to 48 days
Description: Included all participants received at least one dose of glucagon.
Arm/Group | Nasal Glucagon (NG) | Intramuscular (IM) Glucagon
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 44/77 | 35/76
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Nasal Glucagon (NG) (N=77) | Intramuscular (IM) Glucagon (N=76)
Abdominal discomfort (Gastrointestinal disorders) | 1 | 1
Nausea (Gastrointestinal disorders) | 17 | 21
Vomiting (Gastrointestinal disorders) | 13 | 9
Ear pain (Ear and labyrinth disorders) | 2 | 1
Eye pain (Eye disorders) | 1 | 0
Facial pain (General disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 | 1
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 8 | 0
Nasal edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 1
Fatigue (General disorders) | 6 | 5
Lethargy (General disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 | 0
Eye pruritus (Eye disorders) | 2 | 1
Lacrimation increased (Eye disorders) | 7 | 1
Ocular hyperemia (Eye disorders) | 1 | 0
Confusional state (Psychiatric disorders) | 1 | 0
Disturbance in attention (Psychiatric disorders) | 1 | 0
Somnolence (General disorders) | 2 | 0
Hot flush (Nervous system disorders) | 0 | 1
Hyperhidrosis (Nervous system disorders) | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Upper airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 1
Hyperglycemia (Endocrine disorders) | 1 | 0
Anxiety (Psychiatric disorders) | 1 | 0
Headache (Musculoskeletal and connective tissue disorders) | 18 | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No